CLINICAL TRIAL: NCT05199545
Title: Efficacy Study in Phytotherapy of an Association of Plants in the Improvement of Psychological Well-being
Acronym: ROSADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larena SAS (Industry)
Collaborators: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PiL-Clin-ROSADE-021
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Psychological Well-being
MeSH Terms: conditions — Psychological Well-Being | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dietary supplement group (Experimental): 2 tablets / day for 6 weeks of the dietary supplement (Rhodiola rosea L. and Crocus sativus L.), to be taken every day in the morning with a large glass of water, from D1 to D42.
  Interventions: Dietary Supplement: Dietary supplement
- Placebo group (Placebo Comparator): 2 tablets / day for 6 weeks of the placebo, to be taken every day in the morning with a large glass of water, from D1 to D42.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Dietary supplement — Dietary supplement under study is based on Rhodiola rosea L. and Crocus sativus L. extracts
  Arms: Dietary supplement group
Other: Placebo — Placebo of the dietary supplement
  Arms: Placebo group

SUMMARY:
The objective of the study is to compare the effect of a 6-week supplementation with a dietary supplement based on plant extracts to the effect of placebo, in patients with a moderate depressive episode (F32.1 by ICD10 definition) and with moderate symptoms (score HAM-D ≥ 16 and ≤ 23).

DETAILED DESCRIPTION:
Longitudinal, comparative, randomized, placebo-controlled interventional study in 2 parallel groups, double-blind, monocentre, aimed at demonstrating the superiority of the combination of plants over placebo on depressive symptoms.

Each patient will be followed for a maximum of 6 weeks, with 3 visits to the doctor.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 75 years old ;
* Patient with a moderate depressive episode (F32.1 by ICD10 definition) ;
* Score HAM-D ≥ 16 and ≤ 23 at inclusion, corresponding to moderate symptoms ;
* Recent depression (less than 6 months), not managed by antidepressant or psychotherapeutic treatment ;
* Depressive disorder not requiring, in the opinion of the investigator, initiation of antidepressant drug therapy ;
* Patient able to understand the study information, read the information leaflet, and willing to sign the consent form ;
* French speaking patient.

Exclusion Criteria:

* Patient with a depressive disorder of another nature or any other mental illness (schizophrenia, bipolarity, alcohol or drug addiction, etc.);
* Patient at risk of suicide (noted by the investigator, or HAM-D item 3 score > 2) or having attempted suicide in the last 5 years;
* Depression felt for more than 6 months ;
* Patient under psychotropic treatment (current or in the month preceding inclusion) (neuroleptic, anxiolytic, hypnotic);
* Patient on beta-blocker therapy ;
* Patient on dialysis ;
* Patient using products containing piperine or St. John's wort, or having a known effect on mood in the last 30 days ;
* Woman who is pregnant or breastfeeding, or has plans to become pregnant in the next 8 weeks ;
* Patient with an allergy or contraindication to one of the components of the product under study (rhodiola or saffron) ;
* Patient unable to understand information related to the study (mental or linguistic disability) ;
* Patient participating or having participated in the previous 3 months in another clinical trial ;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Evolution of depressive symptoms through Hamilton Depression Scale (HAM-D) at the end of the study | 42 days
  Score HAM-D at D42, adjusted to the value at D0 minimum = 0 and maximum = 53 higher score means a worse outcome

SECONDARY OUTCOMES:
Evolution of depressive symptoms through HAM-D during the study | 42 days
  Evolution of score HAM-D between D0, D21 and D42
Evolution of depressive symptoms through HAM-D sub-scores during the study | 42 days
  Evolution of sub-scores HAM-D between D0, D21 and D42
Rate of responding participants (decrease of ≥ 3 points) at D21 | 21 days
  HAM-D score showing a decrease of ≥ 3 points compared to D0
Rate of responding participants (decrease of ≥ 3 points) at D42 | 42 days
  HAM-D score showing a decrease of ≥ 3 points compared to D0
Rate of responding participants (decrease of ≥ 5 points) at D21 | 21 days
  HAM-D score showing a decrease of ≥ 5 points compared to D0
Rate of responding participants (decrease of ≥ 5 points) at D42 | 42 days
  HAM-D score showing a decrease of ≥ 5 points compared to D0
Rate of participants in remission at D21 | 21 days
  score HAM-D ≤ 7
Rate of participants in remission at D42 | 42 days
  score HAM-D ≤ 7
Evolution of depressive symptoms through Hospital Anxiety and Depression Scale - Depression (HADS-D) during the study | 42 days
  Evolution of sub-scores HADS-D between D0, D21 and D42 minimum = 0 and maximum = 21 higher score means a worse outcome
Evolution of depressive symptoms through Hospital Anxiety and Depression Scale - Anxiety (HADS-A) during the study | 42 days
  Evolution of sub-scores HADS-A between D0, D21 and D42 minimum = 0 and maximum = 21 higher score means a worse outcome
Evolution of physician's general impression of the symptoms during the study | 42 days
  Evolution of Clinical Global Impression-Severity (CGI-S) between D0, D21 and D42 minimum = 1 and maximum = 7 higher score means a worse outcome
Evolution of physician's general impression of the symptoms evolution during the study | 42 days
  Evolution of Clinical Global Impression-Improvement (CGI-I) between D0, D21 and D42 minimum = 1 and maximum = 7 higher score means a worse outcome
Evolution of patient's general impression of the symptoms evolution during the study | 42 days
  Evolution of Patient Global Impression-Improvement (PGI-I) between D0, D21 and D42 minimum = 1 and maximum = 7 higher score means a worse outcome
Adverse events | 42 days
  Number and type of adverse events
Evolution of patient's functional disability in his or her professional, social and family life during the study | 42 days
  Evolution of Sheehan Disability Score (SDS) between D0, D21 and D42 minimum = 0 and maximum = 44 higher score means a worse outcome
Patient satisfaction with complementation at D21 | 21 days
  5-point Likert scale (minimum = 1 and maximum = 5) higher score means a better satisfaction
Patient satisfaction with complementation at D42 | 42 days
  5-point Likert scale
Number of intercurrent visits | 42 days
  Number of intercurrent visits
Concomitant drug use | 42 days
  Number and type of concomitant drugs
Compliance at D21 | 21 days
  Counting of therapeutic units at D21
Compliance at D42 | 42 days
  Counting of therapeutic units at D42
Management prescribed or advised at the end of follow-up | 42 days
  Rate of participants on the same dietary supplement, antidepressant medication, other or without treatment at the end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- CICN - Université Catholique de Louvain, Louvain-la-Neuve, Belgium

IPD SHARING:
Plan to Share IPD: No